CLINICAL TRIAL: NCT05378360
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Therapeutic Exploratory, Phase II Clinical Trial for the Efficacy Investigation and Safety Evaluation of DWP708
Brief Title: DWP708 for Treating Epidermal Growth Factor Receptor Inhibitor Related Skin Toxicities
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWP708201
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2022-05

CONDITIONS: Rash Acneiform
MeSH Terms: conditions — Acneiform Eruptions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo of DWP708 (Placebo Comparator): EGF Cream Placebo evenly apply to skin lesion every 12 hr/day
  Interventions: Biological: DWP708
- DWP708 10 ug/g (Experimental): EGF Cream 10 ug/g evenly apply to skin lesion every 12 hr/day
  Interventions: Biological: DWP708
- DWP708 20 ug/g (Experimental): EGF Cream 20 ug/g evenly apply to skin lesion every 12 hr/day
  Interventions: Biological: DWP708
- DWP708 40 ug/g (Experimental): EGF Cream 40 ug/g evenly apply to skin lesion every 12 hr/day
  Interventions: Biological: DWP708

INTERVENTIONS:
Biological: DWP708 — Placebo Comparator: Placebo of DWP708 / BID / up to 28 days Experimental: DWP708 10 ug/g / BID / up to 28 days Experimental: DWP708 20 ug/g / BID / up to 28 days Experimental: DWP708 40 ug/g / BID / up to 28 days
  Other Names: EGF cream

SUMMARY:
A Multi-center, Randomized, Double-blind, Placebo-controlled, Therapeutic Exploratory, Phase II Clinical Trial for the Efficacy Investigation and Safety Evaluation of DWP708 for Treating Rash Acneiform

DETAILED DESCRIPTION:
All the patients had Grade ≥2 ERSEs according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE) v. 5.0

ELIGIBILITY:
Inclusion Criteria:

1. Age: older than 19
2. Eastern Cooperative Oncology Group (ECOG) performance status 0 -2
3. Patients who have Rash acneiform Gr≥2 (NCI CTCAE v5.0)
4. Patients who are currently administering EGFR TKI or EGFR mAb

Exclusion Criteria:

1. Known allergies, hypersensitivity, or intolerance to study drugs, chemotherapy drugs using this clinical trial
2. Patients with a history of topical medication

   * Steroids within 3 days prior to baseline visit
   * Antihistamine, Antipruritic agents, Antibiotics agents within 1 week prior to baseline visit
   * Tacrolimus, Pimecrolimus within 2 weeks prior to baseline visit

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2022-05-02 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
To estimate the response rate of Rash acneiform | Up to 28 days
  The effectiveness of the DWP708 was defined as follows:
  1. Downgraded to more than 2 steps
  2. Downgraded to ≤Grade 1

SECONDARY OUTCOMES:
To evaluate the patients' Quality of Life (QoL) by Skin evaluation method | Up to 56 days
  SKINDEX-16
To estimate the amount of change papule and/or pustule | Up to 56 days
  Region of interest (10 * 10 cm)

CONTACTS AND LOCATIONS:
Overall Officials: Sung Yong Oh, M.D., Principal Investigator — Dong-A University Hospital
Locations (1):
- Dong-A University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No